CLINICAL TRIAL: NCT00391092
Title: A Randomized, Open-label Study to Compare the Effect of First-line Treatment With Avastin in Combination With Herceptin/Docetaxel and Herceptin/Docetaxel Alone on Progression-free Survival in Patients With HER2 Positive Locally Recurrent or Metastatic Breast Cancer.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Herceptin (Trastuzumab)/Docetaxel in Patients With HER2 Positive Metastatic Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20231
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Trastuzumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Docetaxel; Drug: Herceptin
- 2 (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: Herceptin

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv every 3 weeks
  Arms: 1
Drug: Docetaxel — 100mg/m2 iv every 3 weeks
Drug: Herceptin — 8mg/kg iv loading dose, followed by 6mg/kg iv every 3 weeks

SUMMARY:
This 2 arm study will compare the efficacy and safety of Avastin plus Herceptin/docetaxel, versus Herceptin/docetaxel alone, in patients with HER2 positive locally recurrent or metastatic breast cancer who have not received prior chemotherapy for their metastatic disease. Patients will be randomized 1:1 to receive either Avastin (15mg/kg iv q3weeks) + Herceptin (8mg/kg iv loading dose and 6mg/kg iv q3weeks maintenance) + docetaxel (100mg/m2 iv q3weeks) or Herceptin + docetaxel alone. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* HER2 positive breast cancer with locally recurrent or metastatic lesions;
* eligible for chemotherapy;
* baseline LVEF >=50%.

Exclusion Criteria:

* previous chemotherapy for metastatic or locally recurrent breast cancer;
* previous radiotherapy for metastatic breast cancer (except for metastatic bone pain relief);
* other primary tumor within last 5 years, with the exception of basal or squamous skin cancer, or in situ cancer of the cervix;
* clinically significant cardiovascular disease;
* chronic daily treatment with aspirin (>325mg/day) or clopidogrel (>75mg/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2006-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (83):
- Argentina (8):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mar del Plata
  - Mendoza
  - Salta
  - San Martín
  - Santa Fe
- Australia (10):
  - Lismore, New South Wales
  - Newcastle, New South Wales
  - Port Macquarie, New South Wales
  - Wahroonga, New South Wales
  - Wollongong, New South Wales
  - Auchenflower, Queensland
  - Nambour, Queensland
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Perth, Western Australia
- Austria (4):
  - Graz
  - Salzburg
  - Vienna
  - Vöcklabruck
- Bosnia and Herzegovina (3):
  - Banja Luka
  - Sarajevo
  - Tuzla
- Brazil (5):
  - Goiânia, Goiás
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Barretos, São Paulo
  - São Paulo, São Paulo
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Prague, Czechia
- France (9):
  - Avignon
  - Besançon
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Montpellier
  - Villejuif
- Italy (4):
  - Parma, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Pavia, Lombardy
- Mexico (5):
  - Acapulco
  - Guadalajara
  - Mérida
  - Monterrey
  - Torreón
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (6):
  - Kazan'
  - Moscow
  - Obninsk
  - Ryazan
  - Saint Petersburg
  - Ufa
- Spain (5):
  - Barcelona, Barcelona
  - Sabadell, Barcelona, Barcelona
  - Córdoba, Cordoba
  - Madrid, Madrid
  - Zaragoza, Zaragoza
- Turkey (Türkiye) (2):
  - Izmir
  - Sıhhiye, Ankara
- United Kingdom (8):
  - Exeter
  - London
  - Manchester
  - Nottingham
  - Preston
  - Rhyl
  - Stoke-on-Trent
  - Weston-super-Mare
- Montevideo, Uruguay

REFERENCES:
- [Derived] Gianni L, Romieu GH, Lichinitser M, Serrano SV, Mansutti M, Pivot X, Mariani P, Andre F, Chan A, Lipatov O, Chan S, Wardley A, Greil R, Moore N, Prot S, Pallaud C, Semiglazov V. AVEREL: a randomized phase III Trial evaluating bevacizumab in combination with docetaxel and trastuzumab as first-line therapy for HER2-positive locally recurrent/metastatic breast cancer. J Clin Oncol. 2013 May 10;31(14):1719-25. doi: 10.1200/JCO.2012.44.7912. Epub 2013 Apr 8. PMID 23569311

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participants were randomized 1:1 using a block design randomization procedure with stratification (for prior adjuvant/neo-adjuvant taxane, trastuzumab as part of adjuvant treatment versus no trastuzumab, estrogen/progesterone receptor hormone receptor status and measurable disease) to avoid an imbalance of important prognostic factors.
Groups:
- Trastuzumab + Docetaxel: Trastuzumab 8 milligrams per kilogram (mg/kg) loading dose administered intravenously on Day 1 of Cycle 1, followed by docetaxel 100 milligrams per square meter (mg/m^2) on Day 2 of Cycle 1. Then a maintenance dose of trastuzumab at 6 mg/kg and docetaxel at 100 mg/m^2 were administered intravenously on Day 1 of each 3-weekly cycle until disease progression, unacceptable toxicity (requiring discontinuation of study treatment), or withdrawal of participant's consent, and for a minimum of 6 cycles, respectively.
- Trastuzumab + Bevacizumab + Docetaxel: Trastuzumab 8 mg/kg loading dose administered intravenously on Day 1 of Cycle 1, followed by bevacizumab 15 mg/kg and docetaxel 100 mg/m^2 on Day 2 of Cycle 1. Then a maintenance dose of trastuzumab at 6 mg/kg, bevacizumab 15 mg/kg and docetaxel at 100 mg/m^2 were administered intravenously on Day 1 of each 3-weekly cycle until disease progression, unacceptable toxicity (requiring discontinuation of study treatment), or withdrawal of participant's consent.
Period: Overall Study
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Started | 208 | 216
Received Treatment | 206 | 215
Completed | 0 (This was using a data cutoff of 30 June 2011.) | 0 (This was using a data cutoff of 30 June 2011.)
Not Completed | 208 | 216
Not completed — Death | 78 | 81
Not completed — Lost to Follow-up | 13 | 18
Not completed — Alive on treatment | 29 | 33
Not completed — Alive in follow-up | 88 | 84

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomized participants, regardless of whether they actually received study treatment or not.
Groups:
- Trastuzumab + Docetaxel: Trastuzumab 8 mg/kg loading dose administered intravenously on Day 1 of Cycle 1, followed by docetaxel 100 mg/m^2 on Day 2 of Cycle 1. Then a maintenance dose of trastuzumab at 6 mg/kg and docetaxel at 100 mg/m^2 were administered intravenously on Day 1 of each 3-weekly cycle until disease progression, unacceptable toxicity (requiring discontinuation of study treatment), or withdrawal of participant's consent, and for a minimum of 6 cycles, respectively.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel | Total
Number analyzed (Participants) | 208 | 216 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.71) | 53.5 (10.90) | 53.7 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 216 | 424
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to time of first documented disease progression (unequivocal progression of existing non-target lesions) or death, whichever occurred first as assessed by Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0). Progressive disease is defined using RECIST v1.0 as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started. Primary PFS variable was defined based on the investigators' assessments and the statistical conclusions on the primary efficacy endpoint were based on investigator assessed PFS. PFS was estimated using Kaplan-Meier methods.
Time Frame: Every 9 weeks up to Week 36, thereafter every 12 weeks until disease progression (up to the clinical cutoff of 30 June 2011, up to 4.75 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 208 | 216
months | 13.7 [11.4 to 16.3] | 16.5 [14.1 to 19.1]
Statistical Analysis 1: Comparison: Trastuzumab + Docetaxel vs Trastuzumab + Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.0775, Log Rank (unstratified); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.02]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death, regardless of the cause of death. OS was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 208 | 216
months | 38.3 [34.3 to NA] — The upper range of 95% confidence interval (CI) was not calculable due to immature OS data as greater than 50% of participants were censored at the time of clinical cutoff (30 June 2011). | 38.5 [32.1 to NA] — The upper range of 95% confidence interval (CI) was not calculable due to immature OS data as greater than 50% of participants were censored at the time of clinical cutoff (30 June 2011).
Statistical Analysis 1: Comparison: Trastuzumab + Docetaxel vs Trastuzumab + Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.9543, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.74 to 1.38]

3. Secondary Outcome: Percentage of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Partial Response (PR) in Participants With Measurable Disease at Baseline
Description: Best OR was assessed using RECIST v1.0 criteria. Participants were classified as responders if their best OR was either confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of the longest diameter [LD] of target lesions, taking as reference the baseline sum LD). Participants without any post-baseline assessments were regarded as non-responders. The 95% CI for the one sample binomial using Pearson-Clopper method.
Time Frame: as for outcome 1
Population: ITT Population; only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 176 | 183
percentage of participants | 69.9 [62.5 to 76.6] | 74.3 [67.4 to 80.5]
Statistical Analysis 1: Comparison: Trastuzumab + Docetaxel vs Trastuzumab + Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.3492, Chi-squared; Difference in Response rates = 4.43, 95% CI 2-sided [-5.2 to 14.0] — 95% CI for the difference in response rates using Hauck-Anderson method

4. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time when response (CR or PR per RECIST v1.0) was first documented to the date of disease progression per RECIST v1.0 (unequivocal progression of existing non-target lesions) or death. Progressive disease is defined using RECIST v1.0 as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started.
Time Frame: as for outcome 1
Population: ITT Population: only participants with a best OR of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 123 | 136
months | 11.4 [9.1 to 13.2] | 14.6 [12.0 to 17.1]
Statistical Analysis 1: Comparison: Trastuzumab + Docetaxel vs Trastuzumab + Bevacizumab + Docetaxel; Test type: Superiority or Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.56 to 0.98]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time between randomization and date of disease progression (per RECIST v1.0; unequivocal progression of existing non-target lesions), death, or withdrawal of treatment due to adverse events, withdrawal of informed consent, insufficient therapeutic response, refusal of treatment/failure to co-operate, or failure to return, whichever occurred first. Progressive disease is defined using RECIST v1.0 as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 208 | 216
months | 7.7 [6.3 to 8.6] | 9.8 [7.9 to 10.9]
Statistical Analysis 1: Comparison: Trastuzumab + Docetaxel vs Trastuzumab + Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.5392, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.15]

6. Secondary Outcome: Functional Assessment of Cancer Therapy - Generic (FACT-G) and Functional Assessment of Cancer Therapy - Breast (FACT-B) Subscale Scores
Description: FACT-G is core questionnaire of Functional Assessment of Chronic Illness Therapy (FACIT) measurement system to evaluate quality of life (QoL) in cancer population. FACT-G consisted of 27 questions grouped in 4 domains of general Health-Related QoL (HRQoL): Physical Well-being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB) and Functional Well-Being (FWB); each ranged from 0 (not at all) to 4 (very much). FACT-G ranged between 0-108. Since questions could be reversed coded, as appropriate, before calculating FACT-G, 0 and 108 could be considered worst and best health states. FACT -B is used for assessment of HRQoL in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: 7 items for each physical, functional, social/family; all 3 ranged from 0-28, emotional (6 items) ranged from 0-24, and breast cancer subscale (9 items) ranged from 0-36. All single-item measures ranges from 0-144. High scale score represents a better QoL.
Time Frame: Baseline, Cycles 3, 5, 11, and post progressive disease (PD; 14 to 28 days after disease progression [up to the clinical cutoff of 30 June 2011, up to 4.75 years])
Population: ITT Population; n (number) = number of participants assessed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 173 | 189
units on a scale
  Physical Well-Being: Baseline (n=173,189) | 21.20 (5.74) | 21.47 (5.07)
  Social Well-Being: Baseline (n=173,189) | 20.59 (5.75) | 20.88 (5.77)
  Emotional Well-Being: Baseline (n=173,189) | 14.95 (4.95) | 15.54 (4.44)
  Functional Well-Being: Baseline (n=173,189) | 16.34 (5.83) | 16.36 (5.57)
  Total FACT-G Score: Baseline (n=173,189) | 73.30 (16.60) | 74.49 (14.50)
  Breast Specific: Baseline (n=173,189) | 21.67 (6.43) | 22.84 (5.85)
  Total FACT-B Score: Baseline (n=173,189) | 94.97 (20.50) | 97.46 (17.71)
  Trial Outcome Index: Baseline (n=173,189) | 59.54 (14.03) | 60.85 (12.61)
  Physical Well-Being: Cycle 3 (n=145,173) | 20.19 (4.89) | 19.96 (5.05)
  Social Well-Being: Cycle 3 (n=145,173) | 20.64 (5.32) | 21.19 (5.44)
  Emotional Well-Being: Cycle 3 (n=145,173) | 16.47 (4.19) | 16.70 (4.36)
  Functional Well-Being: Cycle 3 (n=145, 173) | 15.43 (5.33) | 16.20 (5.22)
  Total FACT-G Score: Cycle 3 (n=145,173) | 72.94 (14.81) | 74.05 (14.35)
  Breast Specific: Cycle 3 (n=145,173) | 22.29 (5.78) | 23.17 (5.34)
  Total FACT-B Score: Cycle 3 (n=145,173) | 95.26 (18.52) | 97.23 (17.81)
  Trial Outcome Index: Cycle 3 (n=145,173) | 58.04 (12.80) | 59.33 (12.49)
  Physical Well-Being: Cycle 5 (n=139, 166) | 19.51 (4.83) | 19.67 (4.56)
  Social Well-Being: Cycle 5 (n=139, 166) | 19.36 (5.26) | 20.68 (4.92)
  Emotional Well-Being: Cycle 5 (n=139, 166) | 16.05 (4.44) | 17.07 (4.30)
  Functional Well-Being: Cycle 5 (n=139, 166) | 14.81 (5.45) | 15.78 (4.77)
  Total FACT-G Score: Cycle 5 (n=139, 166) | 69.78 (15.04) | 73.21 (12.49)
  Breast Specific: Cycle 5 (n=139, 166) | 21.65 (5.83) | 23.15 (4.90)
  Total FACT-B Score: Cycle 5 (n=139, 166) | 91.43 (18.81) | 96.36 (15.63)
  Trial Outcome Index: Cycle 5 (n=139, 166) | 55.99 (13.09) | 58.59 (11.01)
  Physical Well-Being: Cycle 11 (n=100, 133) | 21.71 (4.54) | 21.56 (4.53)
  Social Well-Being: Cycle 11 (n=100, 133) | 19.71 (5.74) | 20.78 (4.92)
  Emotional Well-Being: Cycle 11 (n=100, 133) | 15.96 (4.50) | 17.46 (3.70)
  Functional Well-Being: Cycle 11 (n=100, 133) | 16.25 (5.16) | 16.98 (4.92)
  Total FACT-G Score: Cycle 11 (n=100, 133) | 73.26 (15.24) | 76.55 (13.56)
  Breast Specific: Cycle 11 (n=100, 133) | 21.29 (5.55) | 23.80 (4.92)
  Total FACT-B Score: Cycle 11 (n=100, 133) | 94.57 (18.58) | 100.43 (16.97)
  Trial Outcome Index: Cycle 11 (n=100, 133) | 59.19 (12.00) | 62.34 (11.79)
  Physical Well-Being: Post PD (n=33, 39) | 19.94 (4.99) | 20.35 (5.37)
  Social Well-Being: Post PD (n=33, 39) | 19.02 (5.61) | 19.68 (4.77)
  Emotional Well-Being: Post PD (n=33, 39) | 14.76 (4.83) | 14.77 (4.64)
  Functional Well-Being: Post PD (n=33, 39) | 14.13 (5.57) | 15.08 (5.16)
  Total FACT-G Score: Post PD (n=33, 39) | 67.84 (14.21) | 70.04 (15.08)
  Breast Specific: Post PD (n=33, 39) | 22.90 (4.48) | 22.87 (5.14)
  Total FACT-B Score: Post PD (n=33, 39) | 90.74 (16.59) | 92.92 (18.47)
  Trial Outcome Index: Post PD (n=33, 39) | 56.97 (11.16) | 58.47 (12.43)

7. Secondary Outcome: Change From Baseline for FACT-G and FACT-B
Description: as for outcome 6
Time Frame: Baseline, Cycles 3, 5, 11, and post PD (14 to 28 days after disease progression [up to the clinical cutoff of 30 June 2011, up to 4.75 years])
Population: ITT Population; n (number) = number of participants assessed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Number analyzed (Participants) | 145 | 173
units on a scale
  Physical Well-Being: Cycle 3 (n=145,173) | -1.01 (7.54) | -1.51 (7.16)
  Social Well-Being: Cycle 3 (n=145,173) | 0.05 (7.83) | 0.32 (7.93)
  Emotional Well-Being: Cycle 3 (n=145,173) | 1.52 (6.49) | 1.16 (6.22)
  Functional Well-Being: Cycle 3 (n=145, 173) | -0.91 (7.90) | -0.16 (7.63)
  Total FACT-G Score: Cycle 3 (n=145,173) | -0.36 (22.25) | -0.44 (20.40)
  Breast Specific: Cycle 3 (n=145,173) | 0.61 (8.65) | 0.34 (7.92)
  Total FACT-B Score: Cycle 3 (n=145,173) | 0.29 (27.63) | -0.24 (25.12)
  Trial Outcome Index: Cycle 3 (n=145,173) | -1.50 (18.99) | -1.52 (17.75)
  Physical Well-Being: Cycle 5 (n=139, 166) | -1.69 (7.50) | -1.80 (6.82)
  Social Well-Being: Cycle 5 (n=139, 166) | -1.23 (7.79) | -0.20 (7.58)
  Emotional Well-Being: Cycle 5 (n=139, 166) | 1.09 (6.65) | 1.53 (6.18)
  Functional Well-Being: Cycle 5 (n=139, 166) | -1.53 (7.98) | -0.58 (7.33)
  Total FACT-G Score: Cycle 5 (n=139, 166) | -3.53 (22.40) | -1.28 (19.14)
  Breast Specific: Cycle 5 (n=139, 166) | -0.03 (8.68) | 0.31 (7.63)
  Total FACT-B Score: Cycle 5 (n=139, 166) | -3.55 (27.82) | -1.10 (23.62)
  Trial Outcome Index: Cycle 5 (n=139, 166) | -3.55 (19.19) | -2.26 (16.74)
  Physical Well-Being: Cycle 11 (n=100, 133) | 0.51 (7.32) | 0.09 (6.80)
  Social Well-Being: Cycle 11 (n=100, 133) | -0.89 (8.13) | -0.10 (7.58)
  Emotional Well-Being: Cycle 11 (n=100, 133) | 1.00 (6.69) | 1.92 (5.78)
  Functional Well-Being: Cycle 11 (n=100, 133) | -0.09 (7.79) | 0.62 (7.43)
  Total FACT-G Score: Cycle 11 (n=100, 133) | -0.05 (22.54) | 2.06 (19.85)
  Breast Specific: Cycle 11 (n=100, 133) | -0.38 (8.49) | 0.96 (7.64)
  Total FACT-B Score: Cycle 11 (n=100, 133) | -0.41 (27.67) | 2.97 (24.53)
  Trial Outcome Index: Cycle 11 (n=100, 133) | -0.35 (18.46) | 1.49 (17.26)
  Physical Well-Being: Post PD (n=33, 39) | -1.25 (7.61) | -1.12 (7.39)
  Social Well-Being: Post PD (n=33, 39) | -1.58 (8.03) | -1.19 (7.48)
  Emotional Well-Being: Post PD (n=33, 39) | -0.20 (6.92) | -0.78 (6.42)
  Functional Well-Being: Post PD (n=33, 39) | -2.22 (8.06) | -1.28 (7.59)
  Total FACT-G Score: Post PD (n=33, 39) | -5.46 (21.85) | -4.44 (20.92)
  Breast Specific: Post PD (n=33, 39) | 1.22 (7.84) | 0.03 (7.79)
  Total FACT-B Score: Post PD (n=33, 39) | -4.23 (26.37) | -4.55 (25.59)
  Trial Outcome Index: Post PD (n=33, 39) | -2.57 (17.92) | -2.38 (17.70)

ADVERSE EVENTS:
Time Frame: From time of first drug intake up to 28 days after last dose study treatment (up to 4.75 years).
Description: Safety population included all participants who had received at least 1 dose of the trial medication, whether withdrawn prematurely or not.
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab + Bevacizumab + Docetaxel
Serious Adverse Events (participants affected / at risk) | 63/206 | 72/215
Other Adverse Events (participants affected / at risk) | 198/206 | 202/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Docetaxel (N=206) | Trastuzumab + Bevacizumab + Docetaxel (N=215)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 18
Neutropenia (Blood and lymphatic system disorders) | 9 | 6
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 6
Neutropenic infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 0 | 4
Angina gangrenous (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitus (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Stomatitus (Gastrointestinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral vavle incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Asthenia (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Bartholinitis (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Breast discharge (Reproductive system and breast disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Bipolar I Disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
General physical condition (Investigations) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Docetaxel (N=206) | Trastuzumab + Bevacizumab + Docetaxel (N=215)
Alopecia (Skin and subcutaneous tissue disorders) | 141 | 135
Nail disorder (Skin and subcutaneous tissue disorders) | 59 | 68
Rash (Skin and subcutaneous tissue disorders) | 41 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 28
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 19
Nail toxicity (Skin and subcutaneous tissue disorders) | 24 | 15
Erythema (Skin and subcutaneous tissue disorders) | 12 | 16
Onycholysis (Skin and subcutaneous tissue disorders) | 5 | 16
Diarrhoea (Gastrointestinal disorders) | 85 | 107
Nausea (Gastrointestinal disorders) | 76 | 82
Stomatitis (Gastrointestinal disorders) | 61 | 95
Constipation (Gastrointestinal disorders) | 47 | 54
Vomiting (Gastrointestinal disorders) | 37 | 42
Dyspepsia (Gastrointestinal disorders) | 18 | 34
Abdominal pain upper (Gastrointestinal disorders) | 24 | 23
Abdominal pain (Gastrointestinal disorders) | 15 | 27
Haemorrhoids (Gastrointestinal disorders) | 8 | 22
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 8
Toothache (Gastrointestinal disorders) | 7 | 12
Gingival bleeding (Gastrointestinal disorders) | 1 | 15
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 10
Asthenia (General disorders) | 76 | 75
Fatigue (General disorders) | 48 | 69
Oedema peripheral (General disorders) | 72 | 37
Pyrexia (General disorders) | 41 | 51
Influenza like illness (General disorders) | 18 | 17
Chills (General disorders) | 11 | 15
Spinal pain (General disorders) | 4 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 60 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 63
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 35
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 25 | 23
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 18
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Headache (Nervous system disorders) | 40 | 66
Peripheral sensory neuropathy (Nervous system disorders) | 52 | 46
Dysgeusia (Nervous system disorders) | 32 | 37
Paraesthesia (Nervous system disorders) | 28 | 37
Neuropathy peripheral (Nervous system disorders) | 18 | 22
Dizziness (Nervous system disorders) | 16 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 | 109
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 36
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 | 26
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 26
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Lacrimation increased (Eye disorders) | 59 | 75
Conjuctivitis (Eye disorders) | 9 | 22
Dry eye (Eye disorders) | 6 | 12
Urinary tract infection (Infections and infestations) | 33 | 27
Nasopharyngitis (Infections and infestations) | 20 | 18
Cystitis (Infections and infestations) | 17 | 19
Rhinitis (Infections and infestations) | 16 | 17
Upper respiratory tract infection (Infections and infestations) | 11 | 21
Bronchitis (Infections and infestations) | 15 | 9
Hypertension (Vascular disorders) | 27 | 79
Hot flush (Vascular disorders) | 16 | 12
Lymphoedema (Vascular disorders) | 17 | 8
Flushing (Vascular disorders) | 10 | 12
Neutropenia (Blood and lymphatic system disorders) | 51 | 44
Anaemia (Blood and lymphatic system disorders) | 24 | 16
Insomnia (Psychiatric disorders) | 21 | 19
Anxiety (Psychiatric disorders) | 16 | 12
Depression (Psychiatric disorders) | 15 | 13
Decreased appetite (Metabolism and nutrition disorders) | 25 | 39
Weight decreased (Investigations) | 6 | 20
Weight increased (Investigations) | 13 | 8
Proteinuria (Renal and urinary disorders) | 1 | 22
Dysuria (Renal and urinary disorders) | 7 | 13
Left ventricular dysfunction (Cardiac disorders) | 17 | 24
Hypersensitivity (Immune system disorders) | 14 | 10
Vertigo (Ear and labyrinth disorders) | 13 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.